CLINICAL TRIAL: NCT06279364
Title: A Randomized, Open-Label, Multicenter Phase 3 Study of SKB264 Versus Investigator's Choice Chemotherapy as First-Line Treatment in Patients With Unresectable Recurrent or Metastatic Triple-Negative Breast Cancer
Brief Title: A Study of SKB264 Versus Investigator's Choice Chemotherapy in Patients With Unresectable Recurrent or Metastatic Triple-Negative Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Kelun-Biotech Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sichuan Kelun Pharmaceutical Research Institute Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SKB264-Ⅲ-11
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Paclitaxel; 130-nm albumin-bound paclitaxel; Capecitabine; eribulin; Carboplatin

STUDY DESIGN:
Intervention Model Description: Participants will be randomised in a 1:1 ratio to one of two intervention groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SKB264 (Experimental): Participants will receive SKB264 on Day 1 and Day 15 of each 4-week cycle
  Interventions: Drug: SKB264
- Investigator's choice chemotherapy (Active Comparator): If no prior taxane, or prior taxane in the (neo)adjuvant setting and disease-free interval (DFI) >12 months: paclitaxel or nab-paclitaxel.
  If prior taxane and DFI ≤ 12 months: capecitabine, eribulin. If known BRCA1/2 mutation: carboplatin
  Interventions: Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Capecitabine; Drug: Eribulin; Drug: Carboplatin

INTERVENTIONS:
Drug: SKB264 — IV Infusion
  Arms: SKB264
Drug: Paclitaxel — IV Infusion.
  Arms: Investigator's choice chemotherapy
Drug: Nab-paclitaxel — IV infusion.
  Arms: Investigator's choice chemotherapy
Drug: Capecitabine — Tablet. Oral route of administration.
  Arms: Investigator's choice chemotherapy
Drug: Eribulin — IV infusion.
  Arms: Investigator's choice chemotherapy
Drug: Carboplatin — IV infusion.
  Arms: Investigator's choice chemotherapy

SUMMARY:
The aim of the study is to evaluate the efficacy and safety of SKB264 as first-line treatment for patients with unresectable recurrent or metastatic triple-negative breast cancer (TNBC) whose tumors do not express programmed cell death ligand 1 (PD-L1) or in patients with PD-L1 positive tumors who received prior anti-programmed cell death 1 (PD-1)/PD-L1 inhibitor in early setting

DETAILED DESCRIPTION:
This is a randomized, open-label, multicenter, Phase 3 study to evaluate the efficacy and safety of SKB264 versus investigator's choice chemotherapy as first-line treatment for patients with unresectable recurrent or metastatic TNBC whose tumors do not express PD-L1 or in patients with PD-L1 positive tumors who received prior anti-PD-1/PD-L1 inhibitor in early setting.

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically and/or cytologically confirmed TNBC.
2. De novo metastatic or relapsed ≥ 6 months post completion of treatment with curative intent.
3. No prior systemic anti-cancer therapy for unresectable recurrent or metastatic disease.
4. Participants whose tumours are PD-L1-negative, or participants whose tumors are PD-L1 positive and have relapsed after prior anti-PD-1/PD-L1 inhibitor for early-stage disease.
5. At least one measurable lesion per RECIST v1.1.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 with no worsening within 2 weeks prior to randomization.
7. A life expectancy of at least 3 months.
8. Eligible for the chemotherapy options listed as investigator's choice chemotherapy (paclitaxel, nab-paclitaxel, capecitabine, eribulin, or carboplatin) as assessed by the investigator.
9. Adequate organ and bone marrow function.

Key Exclusion Criteria:

1. Active second malignancy.
2. Uncontrolled or clinical significant cardiovascular disease.
3. History of noninfectious pneumonitis/interstitial lung disease (ILD) that required steroids or has current pneumonitis/ILD.
4. Active infection requiring systemic therapy within 2 weeks of randomization.
5. Active hepatitis B or hepatitis C virus infection.
6. Human immunodeficiency virus (HIV) positive or history of acquired immunodeficiency syndrome (AIDS); known active syphilis infection.
7. Known hypersensitivity to SKB264 or its excipients.
8. Previously received TROP2-targeted therapy or topoisomerase 1 inhibitors.
9. Prior treatment with the same investigator's choice chemotherapy (except taxane).
10. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 524 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Randomization up to approximately 40 months
  OS is defined as the time from randomization until the date of death due to any cause.
Progression Free Survival (PFS) assessed by Blinded Independent Central Review (BICR) | Randomization up to approximately 28 months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on BICR or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Randomization up to approximately 28 months
  ORR is defined as the percentage of patients who achieve complete response(CR) or partial response (PR), as assessed by BICR/investigator per RECIST 1.1
Duration of Response (DoR) | Randomization up to approximately 28 months
  DoR is defined as the time from the date of first documented CR or PR until date of documented disease progression per RECIST 1.1, as assessed by BICR/investigator or death due to any cause, whichever occurs first.
Progression-Free Survival (PFS) assessed by Investigator | Randomization up to approximately 28 months
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on investigator or death due to any cause, whichever occurs first.
Disease control rate (DCR) | Randomization up to approximately 28 months
  DCR is defined as the percentage of patients who achieve CR, PR or stable disease (SD), as assessed by BICR/investigator per RECIST 1.1
Time to Response (TTR) | Randomization up to approximately 28 months
  TTR is defined as the time from the date of randomization until the first documentation of CR or PR as assessed by BICR/investigator per RECIST 1.1.
Adverse events(AEs) and severe adverse events (SAEs) | AEs should be collected from signing the informed consent form (ICF) until 30 days after the last dose
  Incidence and severity of AEs and SAEs, and clinically significant lab abnormalities

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China